CLINICAL TRIAL: NCT02521727
Title: A Prospective Colonoscopic Study to Investigate Risk of Colorectal Neoplasms in First-degree Relatives of Patients With Non-advanced Adenomas (NonAA Study)
Brief Title: To Investigate Risk of Colorectal Neoplasms in First-degree Relatives of Patients With Non-advanced Adenomas
Acronym: NonAA
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Other Study IDs: NonAA
Record Dates: First submitted 2015-08-06; First posted 2015-08-13 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Cancer; Colorectal Adenoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool, colonic mucosa
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- exposed siblings/children: Consecutive subjects with non-advanced adenomas will be identified from the colonoscopy database at Prince of Wales Hospital, Alice Ho Miu Ling Nethersole Hospital, Queen Elizabeth Hospital and the bowel cancer screening center at Siu Lek Yuen. Figure 1 illustrates subject recruitment flow chart. They will be consented to provide details on their number of FDR, their FDR contact details, and cause of death in FDR who are deceased. FDR aged 40 to 70 years of consecutive patients with newly diagnosed non-advanced adenomas confirmed from endoscopy and pathology reports will be contacted via phone and invited for an interview and a colonoscopy.
  COLONOSCOPY With informed consents, experienced colonoscopists (GI physicians, colorectal surgeons) will perform colonoscopy under intravenous sedation, midazolam and pethidine after adequate bowel preparation.
- unexposed siblings/children: Subjects (Control) FDR aged 40 to 70 years of asymptomatic average risk subjects who had undergone a colonoscopy in our bowel cancer screening programme between 2010 and 2014 and found to have a normal colonoscopy will be invited to participate by phone and invitation letters, to attend a health talk and to undergo a colonoscopy.
  Confounding factors including use of drugs (aspirin and non-steroidal anti-inflammatory drugs), lifestyle factors (smoking, and diet questionnaire) and history of medical conditions (obesity with calculation of body mass index, diabetes, history of cardiovascular disease) between cases and controls will be recorded.
  COLONOSCOPY With informed consents, experienced colonoscopists (GI physicians, colorectal surgeons) will perform colonoscopy under intravenous sedation, midazolam and pethidine after adequate bowel preparation.

SUMMARY:
The risk of CRC in families of patients with CRC is well established, but it is less well-defined for families of patients with adenomas. Screening recommendations to families when an index subject has an adenoma on colonoscopy are not clear. Previous studies demonstrating an increased CRC risk in close relatives of subjects with adenomas were mostly limited by the lack of a suitable comparison group, did not offer colonoscopy to all relatives or did not have verification on true status of adenoma history in the relatives. A systematic review has reported that most studies cited for risk of CRC in relatives with adenomas have not addressed the intended question. Currently International guidelines recommended screening colonoscopy in close relatives and at a younger age when there is a proband with an adenoma, however this recommendation has not been fully supported by all societies due to the lack of robust evidence. This gap in knowledge highlights the need of well-designed and adequately powered studies to estimate the risk of colorectal neoplasms in subjects who have first-degree relatives with adenomas.

Up to 30% of average risk asymptomatic individuals 50 years or older will have at least one adenoma. Based on current guidelines, nearly half the population will be counseled to undergo a colonoscopy from 40 years old based on a positive family history of adenoma. This will have enormous burden on the healthcare system if screening is implicated in all these individuals. Secondly, not all adenomas carry the same risk. Large or villous adenomas are associated with a nearly 70% increased risk of CRC in first degree relatives (FDR) whereas small adenomas may be associated with a modest increased risk 19. It is therefore important to determine the risk of colorectal neoplasms in families of subjects with non-advanced adenomas to justify more intensive screening in these individuals. Investigators hypothesize that first-degree relatives of patients with non-advanced adenoma have an increased risk of both CRC and adenomas. Investigators aim to quantify this risk, and to identify other individual patient or neoplasm characteristics that may contribute to this increased risk. In addition, Investigators aim to determine molecular alteration profiles of colonic adenoma in siblings of patients with advanced neoplasm.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer and second leading cause of cancer death worldwide. Based on data from the Hong Kong Cancer Registry in 2012, CRC is the second most common cancer in Hong Kong. It is one of the few cancers for which there are convincing data to support the benefits of screeColorectal cancer (CRC) is the third most common cancer and second leading cause of cancer death worldwide. Based on data from the Hong Kong Cancer Registry in 2012, CRC is the second most common cancer in Hong Kong. It is one of the few cancers for which there are convincing data to support the benefits of screening. Currently the removal of adenomas is the most effective way in reducing cancer incidence and mortality. International guidelines recommend screening for individuals at an average risk of CRC from the age of 50 years.

Up to 30% of average risk asymptomatic individuals 50 years or older will have at least one adenoma. Based on current guidelines, nearly half the population will be counseled to undergo a colonoscopy from 40 years old based on a positive family history of adenoma. This will have enormous burden on the healthcare system if screening is implicated in all these individuals. Secondly, not all adenomas carry the same risk. Large or villous adenomas are associated with a nearly 70% increased risk of CRC in first degree relatives (FDR) whereas small adenomas may be associated with a modest increased risk. It is therefore important to determine the risk of colorectal neoplasms in families of subjects with non-advanced adenomas to justify more intensive screening in these individuals.

The molecular pathways leading to tumour development in familial colorectal neoplasms are likely to be different from sporadic cases. Development of new molecular based methods for early detection, prevention or treatment relies heavily on the understanding of the differences between sporadic and familial neoplasms. Identification of genetic mutations can also improve genetic diagnosis and screening protocol of an at risk population.

Investigators hypothesize that first-degree relatives of patients with non-advanced adenoma have an increased risk of both CRC and adenomas. Investigators aim to quantify this risk, and to identify other individual patient or neoplasm characteristics that may contribute to this increased risk. In addition, Investigators aim to determine molecular alteration profiles of colonic adenoma in siblings of patients with advanced neoplasm.

The risk of CRC in families of patients with CRC is well established, but it is less well-defined for families of patients with adenomas. Screening recommendations to families when an index subject has an adenoma on colonoscopy are not clear. Previous studies demonstrating an increased CRC risk in close relatives of subjects with adenomas were mostly limited by the lack of a suitable comparison group, did not offer colonoscopy to all relatives or did not have verification on true status of adenoma history in the relatives. A systematic review has reported that most studies cited for risk of CRC in relatives with adenomas have not addressed the intended question. Currently International guidelines recommended screening colonoscopy in close relatives and at a younger age when there is a proband with an adenoma, however this recommendation has not been fully supported by all societies due to the lack of robust evidence. This gap in knowledge highlights the need of well-designed and adequately powered studies to estimate the risk of colorectal neoplasms in subjects who have first-degree relatives with adenomas.

ELIGIBILITY:
Inclusion Criteria:

* First-degree relatives (aged 40 to 70 years) of individuals diagnosed with non-advanced adenoma on screening colonoscopy as Cases
* FDR of patients with negative findings on colonoscopy identified during the same study period, who are of the same age group as the studied as Cohort

Exclusion Criteria:

* A FDR history of CRC
* A family history compatible with that of Hereditary Non-polyposis Colon Cancer (HNPCC) based on the Amsterdam criteria
* Known Familial Adenomatous Polyposis (FAP) syndrome
* Patients and siblings with known inflammatory bowel disease
* Undergone colonoscopy examinations in the past 5 years
* Severe cardio-pulmonary or other medical co-morbidities that preclude safe colonoscopic examination
* Pregnancy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: siblings of Hong Kong Chinese patients with advanced neoplasm compared with a sex and age-matched control population
Sampling Method: Non-Probability Sample
Enrollment: 828 (Actual)
Dates: Start 2015-11-26 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
number of participants having advanced neoplasms. | one day
  number of participants having advanced neoplasms, (included size of adenoma ≥1cm or villous structure, or high grade dysplasia as confirmed by histological report)

SECONDARY OUTCOMES:
number of participants having colorectal neoplasms | one day
  number of participants having colorectal neoplasms as confirmed by histological report)
number of participants having advanced neoplasms depending on site of non-advanced adenoma in proband | one day
  number of participants having advanced neoplasms (confirmed by histological report) based on site of non-advanced adenoma in proband
number of participants having advanced neoplasms based on the gender of the proband | one day
  number of participants having advanced neoplasms based on the number of participants having advanced neoplasms (confirmed by histological report) based on the gender of the proband
number of participants having advanced neoplasms based on age of the proband | one day
  number of participants having advanced neoplasms (confirmed by histological report) based on the age of the proband

CONTACTS AND LOCATIONS:
Overall Officials: SIEW C NG, MD, Principal Investigator — CUHK
Locations (2):
- Hong Kong (2):
  - Alice Ho Mel Ling Nethersole Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ng SC, Kyaw MH, Suen BY, Tse YK, Wong MCS, Hui AJ, Tak HY, Lau JYW, Sung JJY, Chan FKL. Prospective colonoscopic study to investigate risk of colorectal neoplasms in first-degree relatives of patients with non-advanced adenomas. Gut. 2020 Feb;69(2):304-310. doi: 10.1136/gutjnl-2018-318117. Epub 2019 Apr 26. PMID 31028155